CLINICAL TRIAL: NCT03830151
Title: Hyperpolarized Pyruvate Imaging of Glioma: Imaging-Pathological Correlation
Brief Title: Hyperpolarized Carbon C 13 Pyruvate in Diagnosing Glioma in Patients With Brain Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-0902; NCI-2019-00007 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0902 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Primary Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (carbon C 13 pyruvate, MRSI) (Experimental): Patients receive hyperpolarized carbon C 13 pyruvate IV over 10-20 seconds and then undergo an MRSI scan.
  Interventions: Drug: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Spectroscopic Imaging

INTERVENTIONS:
Drug: Hyperpolarized Carbon C 13 Pyruvate — Given IV
  Other Names: Hyperpolarized 13C-Pyruvate; Hyperpolarized Pyruvate (13C)
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MRSI
  Other Names: 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; Proton Magnetic Resonance Spectroscopic Imaging

SUMMARY:
This trial studies how an imaging agent, hyperpolarized carbon C 13 pyruvate, works in diagnosing glioma in patients with brain tumors. Giving hyperpolarized carbon C 13 pyruvate before an advanced imaging technique called a magnetic resonance spectroscopic imaging (MRSI) scan may help researchers better diagnose glioma in patients with brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish a clinical infrastructure for performing hyperpolarized carbon C 13 pyruvate (hyperpolarized 13-C-pyruvate) imaging in the human brain at MD Anderson.

SECONDARY OBJECTIVES:

I. To assess the correlation between conversion rate of hyperpolarized pyruvate to lactate (kpl) values and Ki-67 quantitation in the tumor.

II. To compare kpl values between tumor and normal brain within patient. III. To assess the association between kpl values and pathology results, including conventional, diffusion, perfusion, and permeability imaging.

IV. To assess the association between kpl values and magnetic resonance (MR) imaging findings.

V. To assess the association between kpl values and genomic findings, including methylation, ribonucleic acid [RNA], and deoxyribonucleic acid [DNA]).

OUTLINE:

Patients receive hyperpolarized carbon C 13 pyruvate intravenously (IV) over 10-20 seconds and then undergo an MRSI scan.

After completion of study, patients are followed up for 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent will be obtained from each participants including healthy volunteers.
* Healthy volunteers will not have contra-indications to MR scanning, but will otherwise not be subject to other selection criteria.
* All patients will be enrolled in study # 2011-0370, the Stereotactic RadPath trial
* Patient is >18 years old, agrees to participate in the clinical study and to complete all required visits and evaluations. The pediatric population has a different disease profile from the glioma patients we hope to recruit. To reduce heterogeneity in the patient population we will not consider patients younger than 18 for this study.
* Patient is a candidate for cerebral tumor resection with lesion suspected to be or previously biopsy proven to be a primary brain tumor.
* Patient is able to understand and give consent to participation in the study.
* Patient agrees to undergo, prior to the procedure, magnetic resonance imaging (MRI, within 14 days and preferably with 3 days of the planned procedure) with perfusion, diffusion and spectroscopic imaging.
* Patient has a GFR > 60. In patients with moderate renal failure (GFR 30-60), an alternate injection with 2 times half-dose multihance (gadobenate dimeglumine) or gadovist (gadobutrol) will be considered, if a contrast exam is deemed clinically necessary.
* Specifically for this Study: Patient is willing to give signed informed consent for C13-Pyruvate MR Spectroscopy.

Exclusion Criteria:

* Healthy volunteers will be screened using same process but will otherwise not be subject to other selection criteria.
* The patient is found to have unfavorable anatomy to indicate that stereotactic biopsy could not be safely performed.
* Pacemakers, electronic stimulation, metallic foreign bodies and devices and/or other conditions that are not MR safe, which include but are not limited to: • electronically, magnetically, and mechanically activated implants • ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators and cardiac pacemakers • metallic splinters in the eye • ferromagnetic hemostatic clips in the central nervous system (CNS) or body • cochlear implants • other pacemakers, e.g., for the carotid sinus • insulin pumps and nerve stimulators • non-MR safe lead wires • prosthetic heart valves (if dehiscence is suspected) • non-ferromagnetic stapedial implants • pregnancy • claustrophobia that does not readily respond to oral medication
* Prior brain tumor treatment, including surgical resection, radiation therapy or chemotherapy for a primary brain neoplasm. Previous biopsy will not disqualify the patient from participation. Remote history (> 6month) of non-CNS malignancy in remission, without evidence of current/ prior brain metastasis, will also not disqualify patient from participating.
* History of cardiac arrhythmia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful collection of hyperpolarized pyruvate magnetic resonance (MR) (HMR) imaging data | Up to 1 year
  The kpl values will be calculated for each biopsy site, tumor border zone, and the contralateral side.

SECONDARY OUTCOMES:
Ki-67 quantitation | Up to 1 year
  Spearman's rank correlation will be used to assess the association between kpl values and Ki-67 if the samples are assumed to be independent. Otherwise, intraclass correlation coefficient (ICC) of random effects models will be used.
Tumor kpl values | Up to 1 year
  Will compare with normal brain kpl values. Linear mixed models will be used.
Normal brain kpl values | Up to 1 year
  Will compare with tumor kpl values. Linear mixed models will be used.
Pathology results | Up to 1 year
  Correlation with kpl values will be determined through generalized linear mixed models.
MR imaging findings | Up to 1 year
  Correlation with kpl values will be determined through generalized linear mixed models.
Genomic findings | Up to 1 year
  Correlation with kpl values will be determined through generalized linear mixed models.

CONTACTS AND LOCATIONS:
Overall Officials: Dawid Schellingerhout, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org